CLINICAL TRIAL: NCT05403944
Title: Optimizing Clinical Outcomes for Patients with Patellofemoral Pain Using Strength Training Rehabilitation Incorporating Power Exercises
Brief Title: Strength or Power Training for Patellofemoral Pain
Acronym: STRIPE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: University of Central Florida (Other); University of Toledo (Other)
Responsible Party: Principal Investigator, Neal Glaviano, Responsible Party, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR22-0038; OR210126 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Patellofemoral Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): The SOC rehabilitation group will complete three strength sessions a week. All participants will be provided an educational pamphlet and exercises will be divided into four components - hip abductors, hip extensors, core, and quadriceps muscles. The load magnitude for exercises will be between 60-70% of their 1 repetition max (1RM), with 3 sets of 12 repetitions and a 2-3-minute rest between sets. Time under tension will be prescribed as slow to moderate, with a 2-second concentric phase and 2-second eccentric phase for each exercise. Hip abductor, hip extensor, and core exercises will be initiated during week 1 and continued for the 6-week intervention, while quadriceps focused exercises will be introduced in weeks 3-6.
  Interventions: Behavioral: Standard of Care Rehabilitation (SOC)
- Strength Training Rehabilitation Incorporating Power Exercises (STRIPE) (Experimental): Those in the STRIPE group will complete two power and one strength training sessions a week. All participants will be provided an educational pamphlet and exercises will be divided into four components - hip abductors, hip extensors, core, and quadriceps muscles. The load magnitude will be greater than 60% of the 1RM, with the goal of continually loading against heavy resistance. Participants will complete 4 sets of 6 repetitions, with 3-5 minutes of rest between sets. Time under tension will be prescribed as <1 second for the concentric phase and 1 second for the eccentric phase of the exercise. The strength training sessions will adhere to same parameters as the SOC. Hip abductor, hip extensor, and core exercises will be initiated during week 1 and continued for the 6-week intervention, while quadriceps focused exercises will be introduced in weeks 3-6.
  Interventions: Behavioral: Strength Training Rehabilitation Incorporating Power Exercises (STRIPE)

INTERVENTIONS:
Behavioral: Standard of Care Rehabilitation (SOC) — 6 weeks of standard of care rehabilitation will be given designed to target the core, hip, and quadriceps muscles. Each participant will be expected to complete 3 supervised telehealth sessions per week.
  Arms: Standard of Care (SOC)
Behavioral: Strength Training Rehabilitation Incorporating Power Exercises (STRIPE) — 6 weeks of STRIPE rehabilitation will be given designed to target the core, hip, and quadriceps muscles. Each participant will be expected to complete 3 supervised telehealth sessions per week.
  Arms: Strength Training Rehabilitation Incorporating Power Exercises (STRIPE)

SUMMARY:
The objective of this study is to compare a novel 6-week strength training rehabilitation incorporating power exercises (STRIPE) program to a standard of care (SOC) program on short-term and long-term pain, subjective function, patellofemoral pain recurrence rates, and secondary outcomes (hip abduction and extension rate of torque development and single-leg squat kinematics). We hypothesize that participants with patellofemoral pain who complete the STRIPE program will have 1) decreased pain, 2) improved subjective function, 3) reduced patellofemoral pain recurrence rates, 4a) improved hip abduction/extension rate of torque development, and 4b) decreased hip adduction and pelvic drop during a single leg squat compared to participants who complete a SOC rehabilitation program.

DETAILED DESCRIPTION:
The proposed study will compare strength-based exercises, which is the standard of care (SOC), that target the hip abductors, hip extensors, lumbo-pelvic, and quadriceps muscles, to a strength training program that utilized power-based exercises (Strength Training Rehabilitation Incorporating Power Exercises [STRIPE]). Individuals with patellofemoral pain, both within the military and general population, present with long-term pain, decreased subjective function, and high recurrence rates. Our primary outcomes are to determine intervention success with self-reported knee pain, measured by the visual analog scale, subjective function, measured by the anterior knee pain scale, and recurrence rates. Recent evidence suggests that two in every three individuals with patellofemoral pain report symptoms up to two years after seeking care, therefore we will assess patellofemoral pain recurrence rates for two years. Additionally, the proposed interventions target gluteal muscle function, supporting our selection of secondary outcome variables. We will assess rate of torque development, as power-based exercises are recommended to improve muscle capacity, of both the targeted gluteus medius and gluteus maximus. We will also assess frontal plane kinematics, as the gluteal muscles are responsible for controlling pelvic and hip motion during functional tasks.

ELIGIBILITY:
Inclusion Criteria:

* Participants to be between the ages of 18-40 years old.
* Insidious onset of symptoms greater than 3 months.
* Worst pain in the previous month of 3/10 with two of the following tasks: prolonged sitting, jumping, squatting, kneeling, running, and stair ambulation.

Exclusion Criteria:

* Other forms of anterior knee pain (Osgood-Schlatter, tendon pain, bursitis, etc.).
* History of lower extremity surgery.
* History of patella subluxation, meniscal injury or ligamentous instability.
* History of referred pain from the lumbar spine.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in knee pain. | Immediately after the intervention and then 6, 12, 18, and 24 months post-intervention.
  Data are presented as knee pain, assessed on the visual analog scale in centimeters, resulting in a score of 0-10, with 0 representing no pain and 10 being worst pain imaginable. Group means and standard deviations will be reported.
Change in self-reported knee function. | Immediately after the intervention and then 6, 12, 18, and 24 months post-intervention.
  Data are presented as self-reported knee function, assessed by the anterior knee pain scale.
  The scale ranged between 0-100, with 0 indicating complete disability and 100 indicating no disability. Group means and standard deviations will be reported.
Patellofemoral pain recurrence | 6 months post intervention, 12-months post intervention, 18-months post intervention, and 24-months post intervention
  The number of patients who report symptoms of patellofemoral pain
Change in hip rate of torque development | Immediately after the intervention.
  Hip abduction and extension rate of torque development will be assessed with a handheld dynamometer. Data are reported as linear, with higher scores representing a faster ability to develop hip muscle force. Group means and standard deviations will be reported.
Change in hip adduction during a single leg squat | Immediately after the intervention and then 6, 12, 18, and 24 months post-intervention.
  Data are presented as a degree, with a higher number representing a higher amount of hip adduction. Group means and standard deviations will be reported.
Change in pelvic drop during a single leg squat | Immediately after the intervention and then 6, 12, 18, and 24 months post-intervention.
  Data are presented as a degree, with a higher number representing a higher amount of pelvic drop. Group means and standard deviations will be reported.

SECONDARY OUTCOMES:
Change in psychological factors | Immediately after the intervention and then 6, 12, 18, and 24 months post-intervention.
  Psychological factors will be measures with the PROMIS-10, a 10-item general self-reported questionnaire that assess general domains related to physical, mental, and social health, in addition to perceived quality of life. PROMIS-10 scores are standardized to the general population using a "T-Score", which is a score of 50 points and a standard deviation of 10-points. Higher scores on the PROMIS-10 indicate a healthier patient. Group means and standard deviations will be reported.
Change in cognitive factors | Immediately after the intervention and then 6, 12, 18, and 24 months post-intervention.
  Cognitive factors will be assessed with the Fear-Avoidance Belief Questionnaire (FABQ), a dimension specific questionnaire. The FABQ contains two subscales - physical activity section that includes six-items, while the work section includes ten-items. The physical activity subscale score range between 0-24 and the work subscale is scored between 0-42. Higher scores identifying greater fear avoidance beliefs for both physical activity and work subscales. Group means and standard deviations will be reported.
Change in coping strategy | Immediately after the intervention and then 6, 12, 18, and 24 months post-intervention.
  Coping strategies will be assessed with the Pain Self-Efficacy Questionnaire (PSEQ), a dimension specific questionnaire. The PSEQ is a ten-item, dimension specific questionnaire that assesses how confident participants are with performing activities while experiencing pain. Each item is rated on a scale ranging from 0 ("not at all confident") to 6 ("completely confident"). The PSEQ score ranges between 0-60, with a higher score representing higher confidence to function with pain. Group means and standard deviations will be reported.
Change in physical activity | Immediately after the intervention and then 6, 12, 18, and 24 months post-intervention.
  Physical activity will be quantified with the International Physical Activity Questionnaire - Short Form (IPAQ-SF), a dimension specific questionnaire. The IPAQ-SF is a 4-item short form that measures physical activity from the previous 7-days. Questions include the number of days per week the participant engaged in vigorous activities, moderate activities, walking, and sitting, with a follow-up question for each asking for duration of time for each task. Group means and standard deviations will be reported.
Change in self-reported knee function | Immediately after the intervention and then 6, 12, 18, and 24 months post-intervention.
  The Knee Injury and Osteoarthritis Outcome Scale (KOOS) and the PFP subscale (KOOS-PF) will provide region and disease specific data throughout the study. The KOOS measures five separate dimensions; pain, symptoms, activities of daily living function, sports and recreational function, and quality of life. Each of the five domains are scored on a scale between 0-100, with lower scores representing greater impairments in self-reported function. The KOOS-PF subscale is an 11-item region specific questionnaire, ranging from 0-100, with greater scores also reflecting greater function.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Glaviano, PhD, Principal Investigator — University of Connecticut
Locations (3):
- United States (3):
  - University of Connecticut, Storrs, Connecticut
  - University of Central Florida, Orlando, Florida
  - University of Toledo, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: No
IPD data will be available on request after manuscript has been published.

REFERENCES:
- [Derived] Glaviano NR, Mangum LC, Bazett-Jones DM, DiStefano LJ, Toland MD, Boling M. Strength Training Rehabilitation Incorporating Power Exercises (STRIPE) for individuals with patellofemoral pain: a randomised controlled trial protocol. BMJ Open Sport Exerc Med. 2023 Jan 17;9(1):e001482. doi: 10.1136/bmjsem-2022-001482. eCollection 2023. PMID 36684710